CLINICAL TRIAL: NCT03851094
Title: Evaluation of an Incentive-based Intervention to Improve 90-day Adherence in PAP-Naive Patients
Acronym: Project Dahlia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Collaborators: Wellth Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLP-18-08-01
Record Dates: First submitted 2019-02-19; First posted 2019-02-22 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Randomization will consist of an allocation ratio of 2:1 (control:treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (Group A) (No Intervention): Standard of care is dictated by the HME normal practices for new CPAP patients.
- Wellth App (Group B) (Experimental): Intervention is use of the Wellth app during the initial compliance period.
  Interventions: Behavioral: Wellth app

INTERVENTIONS:
Behavioral: Wellth app — The intervention is the use of Restful, the Wellth self-management app. There is no clinical treatment intervention, as all participants will be receiving PAP therapy per standard of care. Restful is a smartphone-based patient engagement tool that utilizes concepts from behavioral economics to help patients improve their adherence to therapy. The intervention includes a financial and social incentive reward program.
  Other Names: Restful
  Arms: Wellth App (Group B)

SUMMARY:
This is a prospective, randomized, open-label study to evaluate effectiveness of applying financial and social incentives via a smartphone-based app in helping participants achieve adherence to PAP therapy.

DETAILED DESCRIPTION:
This is a prospective, randomized, two-arm, open-label study to evaluate effectiveness of applying financial and social incentives via a smartphone-based app in helping participants achieve adherence to therapy. Randomization will include an allocation ratio of 2:1 (control:treatment).

Participants will be recruited based on evidence that they are struggling to achieve adherence to therapy after the first 3 nights of usage. Two 'site to participant' contacts are required during this study. These contacts can either occur at the clinical site or remotely (e.g., by telephone). During the initial contact, their interest in the study and eligibility will be confirmed, then they will be consented, asked to complete the Baseline Questionnaire, and their demographic information will be collected on case report forms (CRFs).

Participants randomized to the intervention (Group B) will be provided with information and assistance in downloading Restful to their smartphone and registering with Wellth.

At the final contact (90 days), the participant will be asked to complete an End of Study Questionnaire and the investigative staff will collect PAP therapy data for the trial period and record it on CRFs. Participants in Group B will have access to the Restful app discontinued. This completes the participant's active participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (≥ 18 years of age)
* New diagnosis of OSA
* Prescribed CPAP or APAP for treatment of OSA
* Prescribed a ResMed flow generator compatible with AirView
* Owns a smart phone and is willing to download an app on their phone
* Willing and able to give informed consent
* Can read and comprehend written and spoken English

Exclusion Criteria:

* Have used PAP therapy in the past
* Have been prescribed bi-level or adaptive servo-ventilation therapy
* Are participating in another app-based research study
* Cannot participate for the full duration of the study (at least 90 days)
* Participants who have a medical history or concurrent illness that the investigator considers sufficiently serious to interfere with the conduct, completion, or results of this study, or constitutes an unacceptable risk to the participant for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Merchant, PhD, Study Director — ResMed
Locations (1):
- Sleep Data, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (Group A): Standard of care procedures for new CPAP patients were followed.
Period: Overall Study
Arm/Group | Standard of Care (Group A) | Wellth App (Group B)
Started | 111 | 55
Completed | 111 | 51
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Participant lost device | 0 | 1
Not completed — Participant returned device | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population is comprised of participants that completed the first questionnaire. Missing data has been excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (Group A) | Wellth App (Group B) | Total
Number analyzed (Participants) | 103 | 50 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing data was not included in this analysis.
  years
    number analyzed (Participants) | 102 | 49 | 151
    (all) | 49.1 (12.2) | 48.6 (11.1) | 48.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 17 | 65
  Male | 55 | 33 | 88
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian or Alaska Native | 0 | 0 | 0
  Race/Ethnicity: Asian | 13 | 4 | 17
  Race/Ethnicity: Black or African American | 5 | 4 | 9
  Race/Ethnicity: Hispanic or Latino | 14 | 6 | 20
  Race/Ethnicity: Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Race/Ethnicity: White | 63 | 30 | 93
  Race/Ethnicity: More than One | 5 | 4 | 9
Perceived Disease Severity [Mean (Standard Deviation); unit: units on a scale] — These scores will be used as moderators of the intervention's effectiveness. The unit for this outcome is units on a scale, from 1 to 7. A higher score would mean increased agreeance with higher perceived disease severity.
  units on a scale | 5.48 (0.99) | 5.33 (1.31) | 5.43 (1.10)
Claustrophobia [Mean (Standard Deviation); unit: units on a scale] — These scores will be used as moderators of the intervention's effectiveness. The unit for this outcome is units on a scale between 1 and 5. A higher score would indicate more anxiety with claustrophobic situations.
  units on a scale
    Swimming, wearing a nose plug | 2.1 (1.3) | 2.0 (1.2) | 2.1 (1.2)
    Catch breath during vigorous exercise | 2.1 (1.0) | 2.1 (1.1) | 2.1 (1.0)
    Bad cold, difficult to breathe through nose | 2.3 (1.1) | 2.2 (1.1) | 2.3 (1.1)
    Wearing a mask | 2.4 (1.2) | 2.1 (1.2) | 2.3 (1.2)
    Snorkeling | 2.0 (1.2) | 2.0 (1.3) | 2.0 (1.2)
    Working under car or sink | 1.8 (0.9) | 1.9 (1.1) | 1.8 (1.0)
    Wearing CPAP mask/being on therapy | 2.3 (0.9) | 2.1 (1.1) | 2.2 (1.0)
Coping Skills [Mean (Standard Deviation); unit: units on a scale] — These scores will be used as moderators of the intervention's effectiveness. The unit for this outcome is points. Score ranges from 1 to 5. A higher score will have more of an influence on the relationship between the primary outcome (mean PAP usage) and the intervention.
  units on a scale | 3.53 (0.46) | 3.29 (0.51) | 3.45 (0.49)
Health Literacy [Mean (Standard Deviation); unit: units on a scale] — These scores will be used as moderators of the intervention's effectiveness. The unit for this outcome is units on a scale, ranging from 1 to 5. A lower score would mean increased health literacy.
  units on a scale | 1.3 (0.6) | 1.4 (0.6) | 1.4 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean PAP Usage at 90 Days
Description: Average nightly CPAP use for the 90 day time frame.
Time Frame: 90 days
Population: All enrolled participants are included.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Standard of Care (Group A): Standard of care procedures for a new CPAP patient were applied.
Arm/Group | Standard of Care (Group A) | Wellth App (Group B)
Number analyzed (Participants) | 111 | 55
hours | 4.67 (2.20) | 4.59 (2.36)

2. Secondary Outcome: % of Participants That Meet Medicare Compliance Standard
Description: Medicare compliance standard is using the PAP therapy for at least 4 hours per day on at least 70% of the days in a consecutive 30-day period any time in the first 90 days of therapy. Those that meet this standard are counted in the results below and divided by all patients.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (Group A) | Wellth App (Group B)
Number analyzed (Participants) | 111 | 55
Participants | 88 | 46

3. Secondary Outcome: Change in ESS Questionnaire Scores
Description: Epworth Sleepiness Scale (ESS) will be administered at baseline and 90 days. The unit for this outcome is points. The total score can range from 0 to 24. A larger change or change that decreases from baseline will represent a better outcome. A smaller change or change that increases from baseline will represent a worse outcome. A higher score indicates worse symptoms.
Time Frame: 90 days
Population: Patient reported outcomes data. If participant did not answer both questionnaires, their data is missing from this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Wellth App (Group B): Wellth app
  Wellth app: The intervention is the use of Restful, the Wellth self-management app. There is no clinical treatment intervention, as all participants will be receiving PAP therapy per standard of care. Restful is a smartphone-based patient engagement tool that utilizes concepts from behavioral economics to help patients improve their adherence to therapy. The intervention includes a financial and social incentive reward program.
Arm/Group | Standard of Care (Group A) | Wellth App (Group B)
Number analyzed (Participants) | 92 | 40
score on a scale | -1.99 (3.75) | -2.63 (3.49)

4. Secondary Outcome: Change in FOSQ-10 Questionnaire Scores
Description: Functional Outcomes of Sleep Questionnaire (FOSQ-10) will be administered at baseline and 90 days. The unit for this outcome is points. The range of scores is 5 to 20. Higher scores indicate better functional status. A larger change or change that decreases from baseline will represent a better outcome. A smaller change or change that increases from baseline will represent a worse outcome.
Time Frame: 90 days
Population: Patient reported outcomes data. Only participants that completed both questionnaires are reported here.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care (Group A) | Wellth App (Group B)
Number analyzed (Participants) | 92 | 40
score on a scale | 0.96 (2.55) | 1.74 (2.50)

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected over 90 days for each participant.
Groups:
- Group A: Control group
  Standard of care procedures for new CPAP patients were followed.
- Group B: Wellth app
  Wellth app: The intervention is the use of Restful, the Wellth self-management app. There is no clinical treatment intervention, as all participants will be receiving PAP therapy per standard of care. Restful is a smartphone-based patient engagement tool that utilizes concepts from behavioral economics to help patients improve their adherence to therapy. The intervention includes a financial and social incentive reward program.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/51
Other Adverse Events (participants affected / at risk) | 0/111 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT03851094/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT03851094/ICF_001.pdf